CLINICAL TRIAL: NCT02937506
Title: Patient Satisfaction With Propofol for Out Patient Colonoscopy: A Prospective, Randomized, Double-Blind Study
Brief Title: Patient Satisfaction With Propofol for Out Patient Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mount Carmel Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 131115-3
Record Dates: First submitted 2016-10-17; First posted 2016-10-18 (Estimated); Results first posted 2017-09-27 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2016-10

CONDITIONS: Colon Cancer; IBS; Polyps
Keywords: propofol; colonoscopy; patient satisfaction
MeSH Terms: conditions — Colonic Neoplasms; Polyps; Patient Satisfaction | interventions — Propofol; Fentanyl; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propofol (Experimental): Patients in the treatment arm will be given propofol only when having a colonoscopy.
  Interventions: Drug: Propofol
- Fentanyl Plus Midazolam Only (Experimental): Patients in the control arm will receive only the standard of care medications, fentanyl and midazolam when having a colonoscopy.
  Interventions: Drug: Fentanyl Plus Midazolam

INTERVENTIONS:
Drug: Propofol — The intervention is to use propofol as anesthesia during a colonoscopy.
  Other Names: Diprivan
  Arms: Propofol
Drug: Fentanyl Plus Midazolam — The control is to use standard of care anesthesia, fentanyl and midazolam, during a colonoscopy.
  Other Names: Sublimaze; Versed
  Arms: Fentanyl Plus Midazolam Only

SUMMARY:
The primary purpose of this study is to determine if patient satisfaction with propofol is better than with non-propofol anesthesia for outpatient colonoscopies.

DETAILED DESCRIPTION:
Outpatient colonoscopies are very common, indicated for various reasons, and are more commonly performed in outpatient surgery or endoscopy centers. There is an increase in the use of propofol for sedation because of the short duration of action and quick turn around time. Propofol has been studied extensively for safety and efficacy but patient satisfaction and preference with use has not been well documented in prospective, randomized setting. In the context of the recent changes in healthcare reimbursement where patient satisfaction is becoming an important metric providing data that could improve patient satisfaction is needed.

Patients who presented for a colonoscopy with the Principal Investigator were approached to participate in the study. After obtaining consent the patients were randomized to anesthesia with propofol or control without propofol per random number tables provided by the statistician. The anesthesiologist or nurse anesthetist were asked to remove the paper with the assignment from the envelope to determine which medications to give the patient. Pre-op, intra-op, and post-op data were collected by registered nurses blinded to the anesthetic. The day one follow-up phone call was made by the resident who was blinded to the anesthetic. Data were collected in the pre-op, intra-op, and post-op areas by the researchers who were blinded to the medications used.

ELIGIBILITY:
Inclusion Criteria:

- Patients having an outpatient colonoscopy

Exclusion Criteria:

- High risk patients (ASA IV & V) who are not candidates for colonoscopy in an outpatient center will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2013-11; Primary Completion 2016-03 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anantha Padmanabhan, MD, Principal Investigator — Mount Carmel Health System
Locations (1):
- Mount Carmel Health System, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Propofol | Fentanyl Plus Midazolam Only
Started | 300 | 300
Completed | 300 | 300
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients scheduled for an outpatient colonoscopy at a single ambulatory surgery center.
Groups:
- Total: Total of all reporting groups
Arm/Group | Propofol | Fentanyl Plus Midazolam Only | Total
Number analyzed (Participants) | 300 | 300 | 600
Age, Continuous [Mean (Standard Deviation); unit: Years] — The age of the participant in completed years.
  Years | 61.4 (9.8) | 61.0 (9.4) | 61.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 147 | 285
  Male | 162 | 153 | 315

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction
Description: Satisfaction assessed using self-developed questionnaire.
Time Frame: Patient satisfaction was assessed the day of the procedure.
Population: Same as enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Propofol | Fentanyl Plus Midazolam Only
Number analyzed (Participants) | 300 | 300
Participants
  Very Satisfied | 259 | 222
  Satisfied | 37 | 66
  Neutral/Less than satisfied | 4 | 12

ADVERSE EVENTS:
Arm/Group | Propofol | Fentanyl Plus Midazolam Only
All-Cause Mortality (participants affected / at risk) | 0/300 | 0/300
Serious Adverse Events (participants affected / at risk) | 0/300 | 0/300
Other Adverse Events (participants affected / at risk) | 7/300 | 17/300
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propofol (N=300) | Fentanyl Plus Midazolam Only (N=300)
Nausea/Emesis (Gastrointestinal disorders) | 7 (300) | 17 (300) — Nausea or vomiting up to 24 hours after colonoscopy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No